CLINICAL TRIAL: NCT06880601
Title: Teclistamab Plus Autologous Lymphocytes Infusion for the Treatment of Relapse/Refractory Multiple Myeloma (TALIM)
Brief Title: Teclistamab Plus Autologous Lymphocyte Infusion (ALI) for the Treatment of R/R Multiple Myeloma
Acronym: TALIM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM0125
Record Dates: First submitted 2025-03-14; First posted 2025-03-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myleoma; Multiple Myeloma in Relapse; Multiple Myeloma Refractory
Keywords: Multiple Myeloma; Relapse; Refractoriness; Teclistamab; Autologous lymphocyte infusion
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of Te and ALI (Experimental): Teclistamab plus autologous lymphocyte infusions
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Participants are planned to receive Te monotherapy during the first 5 cycles of treatment (1 cycle= 28 days) Participants will receive Te sc monotherapy consisting of 2 step-up doses (0.06 and 0.3 mg/kg) followed by a weekly treatment dose of 1.5 mg/kg for the first 2 cycles From cycle 3 Day 1, participants will receive Te sc Q2W at the dose of 3 mg/kg- From cycle 7 Day 1, participants will receive Te sc Q4W at the dose of 3 mg/kg.
  After cycle 5, participants in PR or better will continue treatment with Te in combination with 4 Ali infusions (cycles +6, +9, +12, +15). The four doses of ALI will be administered with increasing dosage during Te treatment as follows:
  * before Te Cycle 6: ALI 10 x 10^6/kg
  * before Te Cycle 9: ALI 20 x 10^6/kg
  * before Te Cycle 12: ALI 30 x 10^6/kg
  * before Te Cycle 15: ALI 40 x 10^6/kg
  Teclistamab single agent will be continued until progression, unacceptable toxicity or patients refusal.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of Teclistamab (Te) and autologous lymphocyte infusions (ALI) in relapse refractory multiple myeloma. The main question it aims to answer is: which is the Duration of response (DoR) with Teclistmab and ALI?

Participants will receive Te for 5 cycles. Participants in PR or better after the first five cycles of Te monotherapy will continue treatment with Te in combination with ALI administration starting from cycle 6

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm, phase II trial designed to evaluate the efficacy and safety of the combination of Te and ALI. This combination will be tested in patients with RRMM who are at least in partial response (PR) according to the IMWG criteria after 5 cycles of treatment with Te single agent.

Participants are planned to receive Te monotherapy during the first five cycles of treatment (1 cycle= 28 days)

After cycle 5:

Participants in PR or better will continue treatment with Te in combination with 4 Q12W ALI administration starting from cycle 6 (cycles +6, +9, +12, +15); Participants with < PR after the first five cycles of Te monotherapy (Minimal Response, Stable Disease) will be allowed to continue treatment with Te monotherapy;

After cycle 15:

Patients with PR or better will continue Te monotherapy up to progressive disease, unacceptable toxicity, patients' refusal Patients with < PR (Minimal Response, Stable Disease) will be allowed to continue treatment with Te monotherapy up to progressive disease, unacceptable toxicity, patients' refusal Patients with progressive disease (PD) will stop Te, go off treatment and will be treated according to investigator choice Final evaluation will be performed after the end of Te cycle 24.

ELIGIBILITY:
Inclusion Criteria:

* • Patient has a confirmed diagnosis of MM according to the WHO 2022 classification (18)

  * Patient age is ≥ 18 years of age
  * Patient has a Relapsed or refractory disease as defined below:

    * Relapsed disease is defined as an initial response to previous treatment, followed by confirmed progressive disease by the International Myeloma Working Group (IMWG) (15) criteria >60 days after cessation of treatment
    * Refractory disease is defined as failure to achieve a response or confirmed progressive disease by IMWG criteria (15) during previous treatment or ≤60 days after cessation of treatment.
  * Previous treatment with 1 or 2 lines of treatment (induction plus autologous stem cell transplant plus consolidation and maintenance has to be considered one single line)
  * Previous triple exposure that included an IMID, a PI, and an anti-CD38 antibody (patients with no response or relapse after front line therapy with Dara-VTD or Dara-VRD are eligible)
  * Progressive active symptomatic disease
  * Patient has measurable disease as defined by any of the following:

    * Serum M-protein level ≥0.5 g/dL; or
    * Urine M-protein level ≥200 mg/24 hours; or
    * Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
  * Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
  * Able to adhere to the study visit schedule and all the other protocol procedures and requirements;
  * Patient has the following laboratory parameters:

    * Total lymphocytes count ≥ 0.3 x 109/L
    * Platelet count > 50 x 109/L unless due to bone marrow involvement by MM
    * Conjugated bilirubin up to 2 x ULN unless due to liver involvement by MM
    * Alkaline phosphatase and transaminases up to 2 x ULN unless due to liver involvement by MM
    * Creatinine clearance ≥ 30 ml/min
  * A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test within 2-7 days prior to C1D1
  * Life expectancy ≥ 2 months
  * Successful collection of at least 100 x 106/kg autologous lymphocytes before starting treatment with Te.
  * Patient understands and voluntarily signs an informed consent form

Exclusion Criteria:

* • Previous treatment with > 2 lines of therapy

  * Patient has active central nervous system involvement with MM
  * Received any prior BCMA-directed therapy
  * Received the following prior antimyeloma therapy, within the specified time frame prior to enrollment:

    * Targeted therapy, epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 21 days or ≥5 half-lives, whichever is less
    * Investigational vaccine within 4 weeks
    * Monoclonal antibody therapy within 21 days
    * Cytotoxic therapy within 21 days
    * PI therapy within 14 days
    * IMiD agent therapy within 14 days
    * Radiotherapy within 14 days or focal radiation within 7 days
  * Gene-modified adoptive cell therapy (eg, chimeric antigen receptor modified T cells, NK cells) within 3 months
  * Stem cell transplant:

    * previous allogeneic stem cell transplant
    * autologous stem cell transplant performed within 12 weeks
  * Patients with plasma cell leukemia (presence of 5% or more plasma cells in conventional peripheral blood smear white blood cell differential count)
  * Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients
  * Any ongoing myelodysplastic syndrome or B-cell malignancy (other than MM)
  * Any history of malignancy, other than MM, which is considered at high risk of recurrence requiring systemic therapy
  * Any active malignancy (ie, progressing or requiring treatment change in the last 24 months) other than MM. The only allowed exceptions are malignancies treated within the last 24 months that are considered cured:

    * Non-muscle invasive bladder cancer (solitary Ta-PUNLMP or low grade, <3 cm, no CIS)
    * Non-melanoma skin cancers treated with curative therapy or localized melanoma treated with curative surgical resection alone
    * Non-invasive cervical cancer
    * Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer (anti-hormonal therapy is permitted)
    * Localized prostate cancer (M0, N0) with a Gleason Score ≤7a, treated locally only (RP/RT/focal treatment)
    * Other malignancy that is considered cured with minimal risk of recurrence in consultation with the treating physician
  * Clinically relevant and active liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
  * Patient has any other concurrent severe and/or uncontrolled medical condition(s) (e.g., uncontrolled diabetes mellitus, uncontrolled hypertension, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), active hemorrhage, psychiatric illness, active or uncontrolled infection that in the investigator opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form
  * Participant had major surgery or had significant traumatic injury within 2 weeks prior to enrollment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study.
  * Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrollment
  * Patient has a known history of HIV seropositivity
  * Seropositive for hepatitis B: defined by a positive test for HbsAg. Participants with resolved infection (ie, participants who are HbsAg negative with antibodies to total anti-HBc with or without the presence of anti-HBs) must be screened using RT-PCR measurement of HBV DNA levels. Participants with a known history of HBV infection must be screened using RT-PCR measurement of HBV DNA levels irrespective of serological results. Those who are RT-PCR positive will be excluded. Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by RT-PCR (see Appendix 12).
  * Active hepatitis C infection as measured by positive HCV-RNA testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV-RNA positive) completed antiviral therapy and has undetectable HCV-RNA 12 weeks following the completion of therapy, the participant is eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of response | 24 months from the beginning of Te monotherapy
  Duration of response is the time interval between the date of confirmed response at cycle 5 and the date of documented disease progression or death from any cause, whichever occurs first. Patients who have not progressed or died at the time of analysis will be censored at the date of their last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Principal Investigator — ASUGI - Azienda Sanitaria Universitaria Giuliano Isontina Ospedale Maggiore, Trieste

IPD SHARING:
Plan to Share IPD: No